CLINICAL TRIAL: NCT02332889
Title: A Phase I/Pilot II Trial Combining Decitabine and Vaccine Therapy for Patients With Relapsed or Refractory Pediatric High Grade Gliomas, Medulloblastomas, and Central Nervous System Primitive Neuroectodermal Tumors (CNS PNETs)
Brief Title: Phase I/II: Decitabine/Vaccine Therapy in Relapsed/Refractory Pediatric High Grade Gliomas/Medulloblastomas/CNS PNETs
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Transition to a different immunotherapy strategy in the future at our institution
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14.0855
Record Dates: First submitted 2014-10-20; First posted 2015-01-07 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Gliomas; Medulloblastoma; Neuroectodermal Tumors, Primitive
MeSH Terms: conditions — Glioma; Medulloblastoma; Neuroectodermal Tumors, Primitive | interventions — Vaccines; Decitabine; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine/Vaccine Therapy (Experimental): Biological/Vaccine: Vaccine (autologous dendritic cells) and Drug: Decitabine and Hiltonol
  Interventions: Biological: Vaccine (autologous dendritic cells); Drug: Decitabine and Hiltonol

INTERVENTIONS:
Biological: Vaccine (autologous dendritic cells) — Prior to vaccination, DC will be thawed, washed once with normal saline containing 1% human serum albumin, and viability will be checked (must be > 70%). Peptide pulsed DC will be placed in 1 ml tuberculin syringe(s) and transferred to the study physician for vaccination
Drug: Decitabine and Hiltonol — Patients will receive DAC at a dose of 10 mg/m2/d intravenously (IV) over one hour on days 1-5 of week 1. Hiltonol will be given intramuscularly at the same site immediately following vaccine

SUMMARY:
The main purpose of this study is to determine the safety of using the combination of decitabine and a cancer vaccine plus Hiltonol. The vaccine will be made from the subject's blood cells and is designed to interact in the subject's body with cells that are programmed to fight specific tumor proteins NY-ESO-1, Melanoma Antigen Gene-A1 (MAGE-A1) and Melanoma Antigen Gene-A3 (MAGE-A3). The decitabine will be given to increase the amount and activity of these cancer proteins on the surface of tumor cells to increase the possibility that the vaccine will stimulate cells to act against the tumor cells. Subjects will be assessed to determine how these tumors respond to the treatment.

DETAILED DESCRIPTION:
One of the challenges of the practical application of immunotherapy for brain tumors is the lack of expression of tumor antigens as well as the down-regulation of Major Histocompatibility Complex (MHC Class I and II ) molecules, which are needed for antigen presentation. Considering the ability of 5-aza-2-deoxycytidine (DAC) to facilitate the expression of cancer/testis (CT) antigens and major histocompatibility complex molecules (MHC) and the fact that it has good blood brain barrier penetration, it is reasonable to test this approach in a vaccine study for patients who have experienced disease recurrence. The use of a combined approach to tumor immunotherapy - antigen upregulation followed by vaccination - has not been studied in this patient population, and there is a strong biologic rationale for this strategy.

Patients with pediatric brain tumors (medulloblastoma, CNS PNET, high grade glioma) who have experienced disease relapse or progressive refractory disease will be eligible. Each cycle will consist of DAC at low dose administered over a 5 day period, followed by two weekly vaccinations consisting of autologous dendritic cells pulsed with pooled, overlapping peptide mixes derived from full-length MAGE-A1, MAGE-A3, and NY-ESO-1. This dose of DAC is lower than all previously reported doses that have been safely administered in adult patients with Myelodysplastic syndromes (MDS) and Acute myeloid leukemia (AML), and was used in a previous protocol for relapsed and refractory pediatric neuroblastoma and sarcomas. A novel way of stimulating CD4 and CD8 antigen specific T cells is to use a dendritic cells (DC) vaccine approach in which the cells are pulsed with overlapping peptides derived from these antigens, so that patients from several different HLA backgrounds can be enrolled. Overlapping peptide mixes derived from full-length NY-ESO-1, MAGE-A1, or MAGE-A3 have been acquired and consists of 15-mers, with 11 amino acid overlap. The number of DC given in our study (8-10 x 106 peptide pulsed DC) is within the range of doses given in previous studies. Vaccinations are spaced at weekly intervals, based on multiple previous studies in which this approach is taken, and the fact that in vitro re-stimulation of cytolytic T lymphocyte (CTL) generally occurs on a weekly basis. Granulocyte-macrophage colony-stimulating factor (GM-CSF) is given days 1 through 5 during vaccine weeks, to minimize leukopenia from DAC and to help facilitate antigen presenting cell function. The adjuvant poly-interstitial Cajal-like cell (ICLC; Hiltonol) will be injected immediately after and adjacent to DC vaccine site to enhance DC maturation. We will accrue 10 patients with relapsed, refractory, or progressive pediatric brain tumors over a 3 year period. Cycles will repeat every five weeks, for two cycles. Patients who do not have disease progression after two cycles may receive an additional two cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

Criteria for enrollment:

* Relapsed medulloblastoma, CNS PNET, or high grade glioma. Confirmatory biopsy is required at time of initial diagnosis.
* Because of rapid clinical progression and decline at time of relapse in patients with grade IV gliomas and diffuse intrinsic pontine gliomas (DIPGs), and the 4-6 weeks required to develop vaccine, patients with these tumors will be eligible to enroll and have DCs harvested and stored at the time of diagnosis, but will not be treated with vaccine until time of relapse.
* Age: Patients must be 2 to 25 years of age.

Criteria for treatment:

* The patient must have experienced relapsed, progressive, or refractory disease.
* The patient may have gross tumor that has been treated with chemotherapy or radiation prior to study treatment.
* The patient must have received standard therapy for their tumor.
* The patient must be at least 90 days from primary radiotherapy.
* Hematologic Function: absolute neutrophil (ANC): 1000/uL; Platelet count: 75,000/uL.
* Renal Function: Creatinine clearance or radioisotope glomerular filtration rate (GFR) 70ml/min/1.73 m2 .
* Cardiac Function: Patient must have normal cardiac function documented by:
* Ejection fraction (>55%) documented by echocardiogram or radionuclide multigated acquisition (MUGA) scan evaluation OR
* Fractional shortening (≥28%) documented by echocardiogram
* Liver Function: Total bilirubin 1.5x normal for age, and serum glutamate pyruvate transaminase (SGPT (ALT)) and serum glutamate oxaloacetate transaminase (SGOT (AST)) 3x normal for age.
* Room air pulse oximetry >94%.
* Male and female sexually active patients of reproductive age who wish to participate must agree to use acceptable contraception.
* Lansky/Karnofsky performance scale > 50, electrocorticogram (ECOG) < or = 2 (Appendix I).

Exclusion Criteria:

* Patient is pregnant.
* Patients with a positive result for any of the following diagnostic tests: Hep B Ag, Hep B Core Ab, Hep C Ab, HIV-1 Ab, HIV-2 Ab, human T-cell leukemia virus (HTLV-1 Ab), HTLV-2 Ab, rapid plasma reagin (RPR).
* Patient has a history of autoimmune disease, specifically inflammatory bowel disease, systemic lupus erythematosis, or rheumatoid arthritis.
* Patient is receiving high doses of systemic corticosteroids or concurrent chemotherapy at the time of beginning study treatment. (Maximum dose of dexamethasone allowed is 0.1mg/kg/day not to exceed 4mg/day.)
* Patient has a known systemic hypersensitivity to DAC, Hiltonol, or any vaccine component.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Lucas, MD, Principal Investigator — University of Louisville
Locations (3):
- United States (3):
  - Pediatric Hematology/Oncology University of Louisville, Louisville, Kentucky
  - University of Louisville, Kosair Children's Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky

REFERENCES:
- [Derived] Lang F, Liu Y, Chou FJ, Yang C. Genotoxic therapy and resistance mechanism in gliomas. Pharmacol Ther. 2021 Dec;228:107922. doi: 10.1016/j.pharmthera.2021.107922. Epub 2021 Jun 23. PMID 34171339

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine/Vaccine Therapy: Biological/Vaccine: Vaccine (autologous dendritic cells) and Drug: Decitabine and Hiltonol
  Vaccine (autologous dendritic cells [DC]): Prior to vaccination, DC will be thawed, washed once with normal saline containing 1% human serum albumin, and viability will be checked (must be > 70%). Peptide pulsed DC will be placed in 1 ml tuberculin syringe(s) and transferred to the study physician for vaccination
  Decitabine and Hiltonol: Patients will receive 5-aza-2-deoxycytidine (DAC) at a dose of 10 mg/m2/d intravenously (IV) over one hour on days 1-5 of week 1. Hiltonol will be given intramuscularly at the same site immediately following vaccine
Period: Overall Study
Arm/Group | Decitabine/Vaccine Therapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine/Vaccine Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tolerability (Number of Participants Without Adverse Events)
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine/Vaccine Therapy
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Arm/Group | Decitabine/Vaccine Therapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine/Vaccine Therapy (N=1)
Progressive disease (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No